CLINICAL TRIAL: NCT05185778
Title: Evaluation of Blood Elements Changes and Different Cytokines in Helminthic and Protozoan Infected Patients in Relation to COVID19 Vaccines.
Brief Title: Parasitism & COVID19 Vaccines: New Challenge.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Hany Mohammed, Principal Investigator, Assiut University
Other Study IDs: parasitism & COVID19 vaccines
Record Dates: First submitted 2022-01-09; First posted 2022-01-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Helminths Infection; Protozoan Infections
MeSH Terms: conditions — Protozoan Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- parasitic infected individuals received COVID-19 vaccine: parasitic infected individuals with helminthic or protozoan who received COVID-19 vaccines of any type
  Interventions: Biological: stool examination, blood sample collected
- parasitic infected individuals not received COVID-19 vaccine: parasitic infected individuals with helminthic or protozoan who don't receive COVID-19 vaccines of any type
  Interventions: Biological: stool examination, blood sample collected

INTERVENTIONS:
Biological: stool examination, blood sample collected — Stool examination macroscopically for consistency, color, and presence of blood and/or mucus and microscopically using the following methods:
  * Saline and iodine wet mount.
  * Formalin-ethyl acetate sedimentation method.
  * Modified Ziehl-Nielsen staining : It was done to all cases with manifestations suggestive of protozoa.
    * Collection of peripheral blood samples for Automated CBC and blood indices evaluation.
    * Molecular detection of inflammatory cytokines level (IFNγ, TNFα) and antiinflammatory cytokines (IL4, IL10) by Real-time PCR(polymerase chain reaction).

SUMMARY:
- Parasitic infection is a serious public health problem throughout the world particularly in developing countries including Egypt. The individuals infected with helminths are responding to the parasite infections by a specific Th2 type innate and adaptive immune responses. The Coronavirus Disease 2019 pandemic has affected over 169 million people and caused the death of millions worldwide. COVID vaccines with up to 95% of efficacy and effectiveness have been developed and approved by the Food and Drug Administration (FDA), USA. Moreover, it's reported that vaccination against COVID may lead to Cytokine Storm Syndrome in some vaccinated people with release of large amounts of cytokines as (IFNγ, IL-12, TNFα).

DETAILED DESCRIPTION:
* Parasitic infection is a serious public health problem throughout the world particularly in developing countries including Egypt.
* Stool examination and CBC(complete blood count) are considered as the most easily, affordable and accessible diagnostic tool to suspect the presence of parasitic infection.
* One of the most important laboratory findings in many helminthic and protozoan infections is the high rate of peripheral blood eosinophilia. Giardia lamblia cause increased number of lymphocytes.
* The individuals infected with helminths are responding to the parasite infections by a specific Th2 type innate and adaptive immune responses. The Th2 pattern cytokines predominate in long-term helminth infected individuals.
* During chronic helminths infection, there is increased production of interleukin-4 (IL-4) and interleukin-10 (IL-10) as anti-inflammatory cytokines, as well as increased activation and expansion of eosinophils, mast cells and basophils.
* In addition, IFNγ have an important inflammatory role in many protozoan parasites as Cryptosporidium, Microsporidia, Entamoeba histolytica.
* The Coronavirus Disease 2019 pandemic has affected over 169 million people and caused the death of millions worldwide. COVID vaccines with up to 95% of efficacy and effectiveness have been developed and approved by the Food and Drug Administration (FDA), USA.
* Moreover, it's reported that vaccination against COVID may lead to Cytokine Storm Syndrome in some vaccinated people with release of large amounts of cytokines as (IFNγ, IL-12, TNFα).

ELIGIBILITY:
Inclusion Criteria:

* Vaccinated and non-vaccinated individuals with COVID-19 vaccines who are known to have different parasitic infections (helminths and protozoan) and admitted to Assiut city hospitals.

Exclusion Criteria:

* Bleeding disorders that may alter CBC results.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Vaccinated and non-vaccinated individuals with COVID-19 vaccines who are known to have different parasitic infections (helminths and protozoan) and admitted to Assiut city hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
-Evaluation of CBC changes associated with some helminths and protozoan infected patients. | 3 years
- Estimation of cytokines level in some helminths and protozoan infected patients. | 3 years
- Correlation of CBC changes and cytokines level with COVID-19 vaccine administration. | 3 years

SECONDARY OUTCOMES:
- study parasitic prevalence in community after COVID changes. | 3 years

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol